CLINICAL TRIAL: NCT02198261
Title: Minoxidil Response Testing in Males With Androgenetic Alopecia
Status: Completed | Type: Observational
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-IVD-MINOXIDIL-003
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Androgenetic Alopecia
Keywords: alopecia; androgenetic alopecia; hair loss; minoxidil; 5% minoxidil foam; male pattern hair loss
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plucked hair follicles with visible bulbs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Predicted as non-responders: Patients that the minoxidil response in-vitro diagnostic kit predicted as non-responders. 5% minoxidil topical foam will be administered to subjects in this group.
  Interventions: Drug: 5% minoxidil topical foam
- Predicted as responders: Patients that the minoxidil response in-vitro diagnostic kit predicted as responders. 5% minoxidil topical foam will be administered to subjects in this group.
  Interventions: Drug: 5% minoxidil topical foam

INTERVENTIONS:
Drug: 5% minoxidil topical foam — 5% minoxidil topical foam
  Other Names: Rogaine 5% minoxidil foam; Regaine 5% minoxidil foam

SUMMARY:
Topical minoxidil is the most common drug used for the treatment of AGA in men. While topical minoxidil exhibits a good safety profile, the efficacy in the overall population remains relatively low i.e., 30-40% re-grow hair. To observe significant improvement in hair growth, minoxidil is typically used twice daily for a period of at least 16 weeks. Due to the significant time commitment and low response rate, a diagnostic test to identify non-responders prior to initiating therapy would be advantageous.

Minoxidil is converted in the scalp to its active form, minoxidil sulfate, by the sulfotransferase enzyme SULT1A1. The enzyme expression is variable among individuals. We have demonstrated in two prior feasibility studies that the SULT1A1 enzyme activity in plucked hair follicles correlates with minoxidil response in the treatment of AGA and thus can server as a predictive biomarker.

Consequently, we developed a minoxidil response in-vitro diagnostic kit intended to identify non-responders prior to initiating therapy with 5% topical minoxidil foam.

The primary purpose of this study is to evaluate the clinical validity of the minoxidil response in-vitro diagnostic kit.

ELIGIBILITY:
Inclusion Criteria:

* Males in overall good health
* Age: 18 to 49
* Diagnosed with male androgenetic alopecia with vertex pattern IIIv, IV, or V on the Norwood Hamilton Scale
* Willing to have a mini dot tattoo placed in the target area of the scalp
* Willing to maintain the same hair style, color, shampoo and hair products use, and approximate hair length throughout the study
* Able to give informed consent
* Able to comply with the study requirements for 16 consecutive weeks

Exclusion Criteria:

* Previous adverse event from topical minoxidil treatment
* Does not use and have not used in the past 6 months anti-androgen therapy such as finasteride
* Does not use and have not used in the past 6 months minoxidil (topical or oral)
* Does not take medication known to cause hair thinning such as Coumadin and anti-depressants/anti-psychotics
* Folliculitis
* Scalp psoriasis
* Seborrheic dermatitis
* Inflammatory scalp conditions such as lichen planopilaris

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Males with androgenetic alopecia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-07; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the minoxidil response in-vitro diagnostic kit to predict at baseline the mean change in non-vellus hair count in the target region | baseline to week 16
Sensitivity and specificity of the minoxidil response in-vitro diagnostic kit to predict at baseline the subjects ratings | baseline to week 16

SECONDARY OUTCOMES:
Sensitivity and specificity of the minoxidil response in-vitro diagnostic kit to predict at baseline the treatment efficacy evaluated by expert panel review of global photographs assessing hair regrowth | baseline to week 16
Sensitivity and specificity of the minoxidil response in-vitro diagnostic kit to predict at baseline the mean change in non-vellus hair diameter in the target region | baseline to week 16
Mean change in minoxidil sulfotransferase activity in plucked hairs as measured by the minoxidil response in-vitro diagnostic kit | baseline to week 16

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Keene, MD, Principal Investigator — Physicians Hair Institute; Flavio Grasso, MD, Principal Investigator — Istituto Medico Tricologico/Studi Life Cronos; Rodney Sinclair, MD, Principal Investigator — Sinclair Dermatology
Locations (5):
- United States (2):
  - Physicians Hair Institute, Tucson, Arizona
  - Tennessee Clinical Research Center, Nashville, Tennessee
- Sinclair Dermatology, East Melbourne, Australia
- LTM Medical College & Hospital, Mumbai, India
- Istituto Medico Tricologico/Studi Life Cronos, Florence, Italy

REFERENCES:
- [Background] Roberts J, Desai N, McCoy J, Goren A. Sulfotransferase activity in plucked hair follicles predicts response to topical minoxidil in the treatment of female androgenetic alopecia. Dermatol Ther. 2014 Jul-Aug;27(4):252-4. doi: 10.1111/dth.12130. Epub 2014 Apr 28. PMID 24773771
- [Background] Goren A, Castano JA, McCoy J, Bermudez F, Lotti T. Novel enzymatic assay predicts minoxidil response in the treatment of androgenetic alopecia. Dermatol Ther. 2014 May-Jun;27(3):171-3. doi: 10.1111/dth.12111. Epub 2013 Nov 27. PMID 24283387
- [Background] Buhl AE, Waldon DJ, Baker CA, Johnson GA. Minoxidil sulfate is the active metabolite that stimulates hair follicles. J Invest Dermatol. 1990 Nov;95(5):553-7. doi: 10.1111/1523-1747.ep12504905. PMID 2230218
- [Background] Messenger AG, Rundegren J. Minoxidil: mechanisms of action on hair growth. Br J Dermatol. 2004 Feb;150(2):186-94. doi: 10.1111/j.1365-2133.2004.05785.x. PMID 14996087